CLINICAL TRIAL: NCT05266014
Title: Phase 1/2, Open-Label, Dose-Finding Followed by 2-Year Extension Study to Evaluate Safety and Tolerability of Tinlarebant in Adolescent Subjects With Stargardt Disease
Brief Title: This is a Dose-finding Study Followed by 2-year Extension Study to Evaluate Safety and Tolerability of Tinlarebant in Adolescent Subjects With Stargardt Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RBP4 Pty Ltd (Industry)
Collaborators: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBS-008-CT02
Record Dates: First submitted 2022-01-26; First posted 2022-03-04 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Stargardt Disease
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- tinlarebant (Experimental): Daily, oral administration of one tinlarebant.
  Interventions: Drug: tinlarebant

INTERVENTIONS:
Drug: tinlarebant — Phase 1b Portion: tinlarebant will be self-administered orally once daily for 2 cycles, 14 days per cycle.
  Phase 2 portion: tinlarebant will be self-administered orally once daily for 24 months.

SUMMARY:
Stargardt disease 1 (STGD1) is the most prevalent form of juvenile macular degeneration. It is caused by a rare, inherited autosomal recessive trait, leading to severe and irreversible blindness by the first or second decade of life. Earlier onset of the disease is related to a rapid vision loss, while patients with a later onset tend to have a better prognosis.

This study will enrol subjects aged 12-18 years old with a confirmed clinical diagnosis of Stargardt disease type 1 (STGD1). This study will include 2 phases, the phase 1b portion is to determine the optimal dose for phase 2 based on the extent of retinol binding protein 4 (RBP4) reduction after 2 cycles of tinlarebant treatment. The phase 2 portion will evaluate the safety and efficacy of a single daily dose of tinlarebant over a 24-month treatment period.

ELIGIBILITY:
Major Inclusion Criteria:

Subject must have clinically diagnosed Stargardt disease with at least one mutation identified in the ABCA4 gene.

Major Exclusion Criteria:

Any ocular disease other than Stargardt disease at baseline that, in the opinion of the PI, would complicate assessment of a treatment effect.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
To evaluate systemic and ocular safety and tolerability of tinlarebant. | From baseline to 24 months
  To evaluate safety and tolerability of daily dosing of tinlarebant assessed by incidence and/or severity of ocular and non-ocular adverse events.
The optimal dose for Phase 2. | Up to 24 months
  To determine optimal dose of tinlarebant administered orally in adolescent patients with Stargardt Disease.

SECONDARY OUTCOMES:
Change in atrophic lesion size. | From baseline to 24 months.
Maximum Plasma Concentration (Cmax) of tinlarebant in plasma. | Up to 24 months
Time to Maximum Plasma Concentration (Tmax) of tinlarebant in plasma. | Up to 24 months
Half-life (t1/2) of tinlarebant in plasma. | Up to 24 months
Time to minimal plasma RBP4 level (Tmin) | Up to 24 months
Minimum concentration of RBP4 (Cmin) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (2):
  - Sydney Children's Hospitals Network, Westmead, New South Wales
  - Lions Eye Institute, Perth, Western Australia
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No